CLINICAL TRIAL: NCT04232683
Title: Preoperative Tamsulosin to Prevent Postoperative Urinary Retention in Females After Surgery For Pelvic Floor Disorders
Brief Title: Preoperative Tamsulosin to Prevent Postoperative Urinary Retention After Surgery For Pelvic Floor Disorders
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Eric Hurtado, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLA 19-073
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Urinary Retention
Keywords: Female Pelvic Floor Disorders; Postoperative Urinary Retention; Tamsulosin
MeSH Terms: conditions — Urinary Retention | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Preoperative Tamsulosin (Experimental): The study group will receive one oral dose .4mg of Tamsulosin prior to surgery.
  Interventions: Drug: Tamsulosin 0.4Mg Capsule
- Preoperative Placebo (Placebo Comparator): The control group will receive one oral dose of placebo pill prior to surgery.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Tamsulosin 0.4Mg Capsule — Tamsulosin given preoperatively to detect if rates of urinary retention after female pelvic floor surgeries are decreased
  Arms: Preoperative Tamsulosin
Drug: Placebo oral tablet — Placebo pill given preoperatively
  Other Names: Preoperative Placebo
  Arms: Preoperative Placebo

SUMMARY:
Our hypothesis is that patients receiving preoperative Tamsulosin will have decrease rates of postoperative urinary retention (POUR) after surgery in females for pelvic floor disorders.

DETAILED DESCRIPTION:
This study is a prospective randomized control trial. Patients undergoing pelvic surgery will randomized into two groups. The study group will receive one oral dose of .4mg of Tamsulosin preoperatively.The control group will receive one placebo pill preoperatively. Success or failure of initial voiding trial in postoperative period will be measured. Patients who fail the voiding trial will be discharged home with Foley catheter as is standard protocol at our institution.

ELIGIBILITY:
Inclusion Criteria:

i. Patient undergoing surgery for prolapse with or without mid-urethral sling procedure.

ii. Specific surgical procedures include all vaginal, laparoscopic and robotic reconstructive or obliterative surgeries including the use of mid-urethral slings

Exclusion Criteria:

i. Diagnosis of urinary retention preoperatively (post void residual >150ml)

ii. Malignancy

iii. History of neurological disease

iv. History of spinal cord injuries

v. Allergy to Tamsulosin

vi. Perioperative complications requiring prolonged postoperative bladder drainage

vii. Incontinence procedures other than mid-urethral slings

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tamsulosin Effect | Up to 4 hours after surgery while patient is in post-anesthesia care unit.
  Assess the effect of Tamsulosin in preventing POUR, defined by failure of initial voiding trial postoperatively.

SECONDARY OUTCOMES:
Postoperative Narcotic Use | Up to 4 hours after surgery while patient is in post-anesthesia care unit.
  Amount of postoperative narcotic use will be tracked to assess if increased narcotic use has an effect on postoperative voiding trial (The amount of narctoic use will be measured in milligrams)
Effect of Tamsulosin on postoperative blood pressure | Up to 4 hours after surgery while patient is in post-anesthesia care unit
  A side effect of Tamsulosin in hypotension, therefore, postoperative blood pressure will be evaluated to see if Tamsulosin had a significant impact on blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No